CLINICAL TRIAL: NCT01906502
Title: A Prospective, Open Label Study to Assess the 24-hour IOP Pattern Recorded With SENSIMED Triggerfish® in a Healthy Population
Brief Title: 24-hour IOP Pattern With SENSIMED Triggerfish® in a Healthy Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sensimed AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TF-1217
Record Dates: First submitted 2013-07-17; First posted 2013-07-24 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Healthy Subject

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device (Experimental): Portable device that monitors the 24-hour IOP pattern by a wireless contact lens sensor (CLS) placed on the eye that sends its signals via an antenna around the orbital cavity to a recorder. Upon completion, the recording can be transmitted to a computer for read-out and visualization.
  Interventions: Device: Sensimed Triggerfish

INTERVENTIONS:
Device: Sensimed Triggerfish

SUMMARY:
A database (Snapfish) has been generated at Sensimed compiling all data acquired up to now on healthy volunteers and patients with glaucoma. However, healthy subjects were much younger than glaucoma patients. Additionally, the number of glaucoma patients in Snapfish database was almost twice higher than the number of healthy subjects. As it is generally accepted that intra ocular pressure (IOP) in the aging population is higher than IOP in young adults it is of interest to evaluate the 24-hour IOP pattern of older healthy subjects. Furthermore, improving our knowledge of the "healthy" 24-hour IOP pattern in comparison to glaucoma profiles would be beneficial for management of glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Subject of Caucasian origin
* Healthy subject without previous ocular disease
* Aged between 40 and 80 years, of either sex
* Not more than 6 diopters spherical equivalent in the study eye
* Having given written informed consent, prior to any investigational procedures

Exclusion Criteria:

* Corneal or conjunctival abnormality precluding contact lens adaptation
* Previous refractive surgery
* Occludable or closed iridocorneal angle
* Sleep apnea syndrome
* Subjects with allergy to corneal anesthetic
* Subjects with contraindications for silicone contact lens wear
* Subjects not able to understand the character and individual consequences of the investigation
* Participation in other clinical research within the last 4 weeks

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2013-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The 24-hour IOP pattern recorded with Sensimed Triggerfish (TF) in healthy subjects, aged between 40 and 80 years Secondary | 24-hour

SECONDARY OUTCOMES:
Diurnal and nocturnal IOP patterns in healthy subjects | 24 hours
Assessment of corneal biomechanical properties in healthy population (if available) | 24 hours
Relationship between the 24-hour IOP pattern monitored by TF and the 24-hour blood pressure pattern in healthy subjects (if available) | 24 hours
Assessment of Safety and tolerability through adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Lusky, MD, Principal Investigator — Rabin Medical Center
Locations (5):
- Israel (5):
  - Meir Medical Center, Kfar Saba
  - The Western Galilee Hospital in Naharya, Naharya
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Sourasky Medical Center, Tel Aviv